CLINICAL TRIAL: NCT02866617
Title: Randomized Controlled Clinical Trial Of Oral Health-Related Quality Of Life In Patients Wearing Vacuum Formed Thermoplastic Retainers Constructed On Conventional Stone Models And On 3D Reconstructed Orthodontic Study Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: PPPC/C1-2015/DGD/12
Record Dates: First submitted 2016-05-08; First posted 2016-08-15 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Quality of Life
Keywords: Quality of Life; Vacuum formed thermoplastic retainer; Orthodontic study model; 3D reconstructed study model

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Conventional (Experimental): T1-T2 : VFR constructed on conventional study model T2-T3 : VFR constructed on 3D reconstructed study model
  Interventions: Device: Vacuum Formed Thermoplastic Retainers Constructed On 3D Reconstructed Orthodontic Study Model
- 3D (Experimental): T1-T2 : VFR constructed on 3D reconstructed study model T2-T3 :VFR constructed on conventional study model
  Interventions: Device: Vacuum Formed Thermoplastic Retainers Constructed On 3D Reconstructed Orthodontic Study Model

INTERVENTIONS:
Device: Vacuum Formed Thermoplastic Retainers Constructed On 3D Reconstructed Orthodontic Study Model

SUMMARY:
In dentistry, 3D printing technology is gaining interest. One of the potential application is to construct appliances on 3D reconstructed study models.

The purpose of this study is to compare vacuum formed thermoplastic orthodontic retainers (VFR) constructed on conventional orthodontic study models and reconstructed 3D study models by assessing the oral health-related quality of life (OHRQoL) instrument, Little's Irregularity Index (LII) and compliance.

DETAILED DESCRIPTION:
Aim:

To compare the impact of 2 types of vacuum formed thermoplastic retainers on patients.

Objectives:

1. To compare oral health-related quality of life in patients wearing vacuum formed thermoplastic retainers constructed on a conventional orthodontic study model and reconstructed 3D study model up to 6 months.
2. To compare compliance between vacuum formed thermoplastic retainers constructed on a conventional orthodontic study model and reconstructed 3D study model up to 6 months.
3. To compare stability in patients wearing vacuum formed thermoplastic retainers constructed on a conventional orthodontic study model and reconstructed 3D study model up to 6 months.

Research Methadology

Ethical Consideration:

Application for ethical approval from Medical Ethics Committee, Faculty of Dentistry, University of Malaya.

Study population

This randomized controlled clinical trial will include existing patients who visited the Faculty of Dentistry, University of Malaya, for fixed orthodontic treatment and are due to have their fixed appliances removed.

5.2 Sample Size Estimation

Sample size estimation is based on previous study done by Jäderberg et al (2012) and calculated using PS Software (Power and Sample Size Calculation).

A sample size calculation was performed based on an alpha significance level of 0.05 and a beta of 0.1 to achieve 90 per cent power to detect a clinically meaningful difference of 1.0 mm [standard deviation (SD) 1.0] between the groups. The sample size calculation revealed that 22 pairs of sample were sufficient. This number of sample size will also achieve a moderate Pearson Product Moment correlation between the two groups. However, to compensate for possible dropouts, 30 pairs were enrolled in this clinical trials.

5.4 Materials and methods

1. Enrollment & Randomization Potential subjects will be recruited from the patients receiving orthodontic treatment at the Faculty of Dentistry, University of Malaya. Patients were screened based on when they were scheduled for debonding and the inclusion and exclusion criteria listed above. An online random number generator was used to create a randomization list of study numbers matched to either Group A or Group B. The day of debonding potential subjects were given consent and officially enrolled in the study.
2. Study Groups As the flow chart below illustrates, two study groups existed for this randomized cross-over observational study. Each study group received 3 sets of vacuum formed thermoplastic retainers. Group A will wear vacuum formed thermoplastic retainers constructed by laboratory technician according to their standard protocol for 1 week from the day of debond, then vacuum formed thermoplastic retainers constructed on stone study model by one dentist after 1 week of debond for 3 months and later vacuum formed thermoplastic retainers constructed on 3D reconstructed study model for another 3 months.

   Group B will wear vacuum formed thermoplastic retainers constructed by laboratory technician according to their standard protocol for 1 week from the day of debond, then vacuum formed thermoplastic retainers constructed on 3D reconstructed study model by one dentist after 1 week of debond for 3 months and later vacuum formed thermoplastic retainers constructed on stone study model for another 3 months.
3. Study Visit #1- Debonding Appointment

   All subjects were debonded by resident doctor, all residual composite removed, and teeth appropriately polished. Final photos were taken per University Clinic protocol. After debond, maxillary and mandibular alginate impressions (Hydrogum 5, Zhermack, Italy) will be obtained from each sample; two for working model and one for study model). One set of impression will be sent to University's Orthodontic Laboratory for construction of vacuum formed thermoplastic retainer by the laboratory technician for 1st appliance (to be issued on the same day of debond). The vacuum formed thermoplastic retainerss were made in the lab using thermoplastic material and clinic's Biostar machine available at the lab using the standard instructions provided by the manufacturer. vacuum formed thermoplastic retainerss were cooled and trimmed accordingly. Clinically vacuum formed thermoplastic retainerss were evaluated by resident doctor intra orally and were adjusted for patient comfort. All subjects were instructed to wear their retainers full time, only remove to eat, brush, and clean. For the remaining two sets of impression, the impression is poured in dental stone within 24hours.
4. Acquisition of stone study model. Impressions obtained will be disinfect before casting. The white stone (Elite Ortho, Zhermack, Italy) is mixed and tapped into the impression a little at a time to ensure no air is trapped within the stone mix and some stone is used to form the base. Once the stone has set sufficiently, the impression is inverted on the base. When casting the lower impression, stone in the lingual section is removed before setting fully to ensure that the impression can easily be removed from the model.

Once the base has fully set the impression will be carefully removed from the stone and gradually lifted from the model using a plaster knife. The resulting stone model is then trimmed using a model trimmer. The base of the model parallel to the occlusal plane is trimmed to ensure even adaption of the thermoforming material. The back edge of the model should be trimmed so that it is at 90° to the sagittal plane. The labial and buccal sides of the model should be trimmed round so that the final model is a 'D' shape.

5 : Acquisition of digital model. Conventional study model will be scanned using structured light scanner (Maestro 3D, Age Solutions, Inc, Italy) via EasyDentalScan software (Age Solutions, Inc) to produce 3D digital model. The scanned data for both upper and lower conventional study models will be saved and exported as binary stereolithographic (.stl) files.

6 : Acquisition of reconstructed model. A Fused Deposition Modelling (FDM) machine (UP! 2 Plus 3D Printer) containing acrylonitrile butadiene styrene (ABS) plastic will be used to construct replica (RP) model from digital file according to manufacturing instructions. This process will be done by CBMTI SDN BHD ( a subsidiary of UM CAPITAL BERHAD), Institute of Postgraduate Studies, University of Malaya.

The prototyping process begins with unwinding the feedstock filament from a reel and feeding it through the liquefier located inside the system working envelop, as shown in figure below, where it gets gradually heated by temperature gradient provided by a number of coils wrapped helically about the axis of the liquefier .

The heated liquefier melts the plastic filament and deposits the melt through a nozzle attached at the exit controlling the diameter of final extrudate. Two step motors at the entrance of liquefier make sure a continuous supply of material during the model build-up. The nozzle and liquefier assembly is mounted onto a mechanical stage numerically controlled in X-Y plane. Upon receipt of precise tool paths prepared by the Insight software, the nozzle moves over the foam substrate depositing a thin bead of thermoplastic model material along with any necessary support structure. Deposition of fine extruded filaments onto the substrate produces a layer corresponding to a slice of the CAD model of the object. Once a layer is built the substrate moves down in z direction in order to prepare the stage for the deposition of next layer. The deposited filaments cool down immediately below the glass transition temperature of the polymer and get hardened. The entire build system is contained within a temperature- controlled environment with temperatures just below the glass-transition temperature of the polymer to provide an efficient intra-layer bonding.

7 : Acquisition of vacuum formed thermoplastic retainer

Each VFR was constructed from an Erkodur blank (Erkodent, Erich Kopp, GmbH, Pfalzgrafenweiler, Germany) 1.5 mm in thickness using the standard instructions provided by the laboratory's Biostar machine.

Retainer Designs:

vacuum formed thermoplastic retainerss Designs- Extraction and Non-extraction Cases

* Upper- Trimmed for 1-2mm of facial gingival coverage, palatal coverage, and 2nd Molar occlusal coverage
* Lower- Trimmed for 1-2mm of facial and lingual gingival coverage, 2nd Molar occlusal coverage.

  8 : T2 and T3 visit: Issuing the vacuum formed thermoplastic retainer. The 2nd retainers will be fitted within 1 week after debond (T1) and the 3rd retainers is fitted 3 months (T2) after debond. The duration of retainer wear was standardized based on the standard protocol for retainer wear in the practice. The patients were instructed to wear the vacuum formed thermoplastic retainers 24 hours a day for the first week and remove them only for eating and brushing their teeth. After the first week, wear time was reduced to 10 hours a day (Thickett and Power, 2009). All patients will be provided with standardized oral and written instructions on how to use the retainers by one dentist.

The subjects were reviewed by a member of the research team at 2 intervals, 3 months (T2) and 6 months (T3) after debond. At the 3 month (T2) review appointment, the subjects will be given the Questionnaire Q2 to be filled up. Later, the 3rd retainer will be given to the subjects and again to be reviewed after 3 months (T3) of 3rd retainer issued ( 6 months after debond) and questionnaire Q3 will be administered.

ELIGIBILITY:
1. Inclusion criteria

   1. fixed appliance treatment following both arches;
   2. indicated for vacuum formed thermoplastic retainers as retention phase in treatment plan;
2. Exclusion criteria:

   1. single-arch or sectional fixed appliance treatment,
   2. hypodontia requiring tooth replacement on the retainer as a temporary measure,
   3. undergone rapid maxillary expansion,
   4. indicated for double retention regime (bonded retainers),
   5. early debonding patients.
   6. patients intending to relocate within the study period
   7. patient with learning difficulties and can't read written instructions/questionnaire in English or Malay
   8. patient with cleft lip or palate
   9. has undergone surgical treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Oral Health-Related Quality Of Life | 6 month

SECONDARY OUTCOMES:
Little's Irregularity Index | 6 month

OTHER OUTCOMES:
Patient's compliance on wearing orthodontic retainers | 6 month
  A survey of patient's compliance wearing the orthodontic retainers in 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wan Nurazreena Wan Hassan, BDS, Principal Investigator — University of Malaya
Locations (1):
- Faculty of Dentistry, University of Malaya, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Mohd Tahir N, Wan Hassan WN, Saub R. Comparing retainers constructed on conventional stone models and on 3D printed models: a randomized crossover clinical study. Eur J Orthod. 2019 Aug 8;41(4):370-380. doi: 10.1093/ejo/cjy063. PMID 30321319